CLINICAL TRIAL: NCT02646956
Title: Taste Preferences for Nutritive and Non Nutritive Sweeteners Among Children and Adults
Acronym: TNNS
Status: Completed | Type: Observational
Sponsor: Monell Chemical Senses Center (Other)
Responsible Party: Sponsor
Other Study IDs: NIH DC011287
Record Dates: First submitted 2015-12-18; First posted 2016-01-06 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2015-12

CONDITIONS: Development
Keywords: Sweet Taste; Psychophysics; Genetics; Diet; Age; Nonnutritive Sweetener
MeSH Terms: interventions — Sweetening Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Salivary samples obtained for genotyping of taste receptor genes
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Age Group-Children: Children between ages of 7 and 14
  Interventions: Other: sweeteners
- Age Group-Adults: Healthy adults who are the parent of the children
  Interventions: Other: sweeteners

INTERVENTIONS:
Other: sweeteners — Participants tasted a variety of nutritive and nonnutritive sweeteners

SUMMARY:
The goal of the study is to determine whether there are age-, diet- and genetically-related differences in the perception of sweeteners, both nutritive and non-nutritive.

DETAILED DESCRIPTION:
This is an observational 3-day study of children between the ages of 7 and 14 and their mothers. A variety of psychophysical methods determined liking for each of the sweeteners and saliva samples were obtained for genotyping of taste receptor genes. Anthropometric and dietary intake measures were also collected.

ELIGIBILITY:
Inclusion Criteria:

* Healthy

Exclusion Criteria:

* Allergies and taking medication that affected taste

Ages: 7 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy children and adults living in the Philadelphia area
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2014-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Liking for the taste of sweeteners measured via the 3-point facial hedonic scale. | Through study completion, an average of 6 months.
Liking for the taste of sweeteners measured via the 5-point facial hedonic scale | Through study completion, an average of 6 months.
Liking for the taste of sweeteners measured via the Monell forced-choice, paired-comparison tracking procedure. | Through study completion, an average of 6 months.

SECONDARY OUTCOMES:
Genotyping of taste receptor genes via saliva donation | Through study completion, an average of 6 months
  Genotyping will be completed to measure associations between individual taste receptor genotypes and liking of sweeteners.
BMI calculated from body weight and height measures | Through study completion, an average of 6 months
  BMI will be calculated to examine associations between this measure and liking for sweeteners.
One day dietary intake collected via the Automated Self-Administered 24-hour dietary recall (ASA24). | Through study completion, an average of 6 months
  Dietary recall will be completed to examine associations between added sugar intake and liking for sweeteners.

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Mennella, PhD, Principal Investigator — Monell Chemical Senses Center

IPD SHARING:
Plan to Share IPD: No